CLINICAL TRIAL: NCT05681702
Title: Tailoring Bleeding Reduction Approaches in Patients Undergoing Percutaneous Coronary Interventions: Comparative Pharmacodynamic Effects of Potent P2Y12 Inhibitor Monotherapy Versus Dual Antiplatelet Therapy De-escalation
Brief Title: Tailoring Bleeding Reduction Approaches in Patients Undergoing PCI
Acronym: TAILOR BLEED
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202202835
Record Dates: First submitted 2023-01-04; First posted 2023-01-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous coronary intervention; Dual antiplatelet therapy; Bleeding
MeSH Terms: conditions — Coronary Artery Disease; Hemorrhage | interventions — Aspirin; Clopidogrel; Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Intervention Model Description: Prospective randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DAPT de-escalation (Active Comparator): Aspirin 81-mg od and clopidogrel 75-mg qd.
  Interventions: Drug: aspirin plus clopidogrel
- Potent P2Y12 monotherapy (Experimental): Potent P2Y12 inhibitor with prasugrel 10 mg od or ticagrelor 90 mg BID.
  Interventions: Drug: prasugrel or ticagrelor

INTERVENTIONS:
Drug: aspirin plus clopidogrel — After at least 30 days of DAPT [with aspirin 81-mg od and a potent P2Y12 inhibitor (prasugrel 10 mg od or ticagrelor 90-mg BID)] in chronic coronary syndrome or after at least 90 days of DAPT in acute coronary syndromes; patients will continue aspirin and switch to clopidogrel 75-mg.
  Arms: DAPT de-escalation
Drug: prasugrel or ticagrelor — After at least 30 days of DAPT [with aspirin 81-mg od and a potent P2Y12 inhibitor (prasugrel 10 mg od or ticagrelor 90-mg BID)] in chronic coronary syndrome or after at least 90 days of DAPT in acute coronary syndromes; patients will drop aspirin and continue prasugrel or ticagrelor.
  Arms: Potent P2Y12 monotherapy

SUMMARY:
Two strategies have both proven to be effective in reducing bleeding complications while preserving efficacy compared with maintaining long-term DAPT with aspirin and a potent P2Y12 inhibitor: a) DAPT de-escalation (i.e., switching from prasugrel or ticagrelor to clopidogrel while maintaining aspirin) and b) potent P2Y12 inhibitor monotherapy (i.e., maintaining prasugrel or ticagrelor and dropping aspirin). These strategies have been tested in a number of trials and have led to changes in practice guidelines to consider either one of these strategies as bleeding reduction approaches among ACS patients undergoing PCI. However, comparative assessments between DAPT de-escalation and potent P2Y12 inhibitor monotherapy are lacking.

DETAILED DESCRIPTION:
Dual antiplatelet therapy (DAPT) with aspirin and a P2Y12 receptor inhibitor represents the standard of care for the prevention of atherothrombotic events in patients with acute coronary syndrome (ACS) or undergoing percutaneous coronary intervention (PCI). In particular, in ACS patients undergoing PCI, DAPT is initiated during the index event and maintained for up to 12 months to prevent stent-related complications as well as ischemic recurrences in non-treated coronary segments. Three oral P2Y12 inhibitors are currently recommended in this setting: clopidogrel, prasugrel, and ticagrelor. However, in ACS patients undergoing PCI, prasugrel and ticagrelor are preferred over clopidogrel based on results of large-scale clinical trials showing their superior reduction in ischemic events, including stent thrombosis. Nevertheless, such ischemic benefit occurs at the expense of increased bleeding. These observations are attributed to the greater antiplatelet potency of prasugrel and ticagrelor over clopidogrel. Importantly, accruing evidence support that bleeding complications carry significant prognostic implications, including increased mortality, underscoring the need to define antiplatelet strategies associated with reduced bleeding while preserving ischemic efficacy. The notion that most recurrent ischemic events, including stent thrombosis, occur early after the index event (i.e., 1-3 months post PCI) has prompted the design of clinical trials assessing antiplatelet treatment regimens consisting in the use of agents with enhanced platelet inhibition during the first months after PCI followed by approaches with reduced platelet inhibition. To this extent, two strategies have both proven to be effective in reducing bleeding complications while preserving efficacy compared with maintaining long-term DAPT with aspirin and a potent P2Y12 inhibitor: a) DAPT de-escalation (i.e., switching from prasugrel or ticagrelor to clopidogrel while maintaining aspirin) and b) potent P2Y12 inhibitor monotherapy (i.e., maintaining prasugrel or ticagrelor and dropping aspirin). These strategies have been tested in a number of trials and have led to changes in practice guidelines to consider either one of these strategies as bleeding reduction approaches among ACS patients undergoing PCI. However, comparative assessments between DAPT de-escalation and potent P2Y12 inhibitor monotherapy are lacking.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who presented with chronic coronary syndrome, underwent PCI and have been on maintenance treatment with DAPT, composed of low-dose aspirin (81mg od) and prasugrel (10 mg od) or ticagrelor (90 mg bid) for at least 30 days. Or patients that presented with an Acute coronary syndrome (ACS) event and underwent PCI and have been on maintenance treatment with DAPT, composed of low-dose aspirin (81mg od) and prasugrel (10mg od) or ticagrelor (90mg bid) for 3 months or greater.
2. Age ≥18 years old
3. Provide written informed consent

Exclusion Criteria:

1. Prior history of stent thrombosis
2. On treatment with any oral anticoagulant (vitamin K antagonists, dabigatran, rivaroxaban, apixaban, edoxaban) or chronic low-molecular-weight heparin (at venous thrombosis treatment, not for prophylaxis)
3. Renal failure requiring dialysis
4. Patients with known bleeding diathesis or coagulation disorders
5. Known severe hepatic impairment
6. Hemodynamic instability
7. Hypersensitivity to clopidogrel
8. Pregnant and breastfeeding women [women of childbearing age must use reliable birth control (i.e., oral contraceptives) while participating in the study]

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Thrombus formation defined as AUC measured by T-TAS | 30 days
  Comparison of the area under the curve (AUC) determined by Total Thrombus formation Analysis System (T-TAS) between potent P2Y12 monotherapy strategy and de-escalation strategy (trough effect).

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD,PhD, Principal Investigator — University of Florida College of Medicine Jacksonville
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capodanno D, Baber U, Bhatt DL, Collet JP, Dangas G, Franchi F, Gibson CM, Gwon HC, Kastrati A, Kimura T, Lemos PA, Lopes RD, Mehran R, O'Donoghue ML, Rao SV, Rollini F, Serruys PW, Steg PG, Storey RF, Valgimigli M, Vranckx P, Watanabe H, Windecker S, Angiolillo DJ. P2Y12 inhibitor monotherapy in patients undergoing percutaneous coronary intervention. Nat Rev Cardiol. 2022 Dec;19(12):829-844. doi: 10.1038/s41569-022-00725-6. Epub 2022 Jun 13. PMID 35697777
- [Background] Capodanno D, Bhatt DL, Gibson CM, James S, Kimura T, Mehran R, Rao SV, Steg PG, Urban P, Valgimigli M, Windecker S, Angiolillo DJ. Bleeding avoidance strategies in percutaneous coronary intervention. Nat Rev Cardiol. 2022 Feb;19(2):117-132. doi: 10.1038/s41569-021-00598-1. Epub 2021 Aug 23. PMID 34426673